CLINICAL TRIAL: NCT03503890
Title: Expanded Access to Rovalpituzumab Tesirine
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C18-915; C19-917 (Other Grant/Funding Number: AbbVie)
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Small Cell Lung Cancer
Keywords: Expanded Access, Pre-approval Access, Compassionate Use, Special Access Program, Named Patient Basis, Special Access Scheme
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — rovalpituzumab tesirine

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: rovalpituzumab tesirine — intravenous
  Other Names: SC16LD6.5

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to Rovalpituzumab Tesirine prior to approval by the local regulatory agency. Availability will depend on territory eligibility. Participating sites will be added as they apply for and are approved for the EAP. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* The participant must not be eligible for a Rovalpituzumab Tesirine clinical trial.
* Pediatric participants may be evaluated on a case by case basis.

Exclusion Criteria:

* None.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie